CLINICAL TRIAL: NCT03548233
Title: BCG Vaccination Scar Formation in Children Under Five Years :Factors Affecting Its Formation and Subsequent Adverse Effects .
Acronym: bcgscars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abd elhamid Mahran, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bcgvaccinationscars
Record Dates: First submitted 2018-05-11; First posted 2018-06-07 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: BCG Vaccination Reaction
MeSH Terms: interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: bcg vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bcg vaccinated (Other): children under five year vaccinated by bcg vaccine
  Interventions: Biological: bcg vaccine

INTERVENTIONS:
Biological: bcg vaccine — live attenuated vaccine

SUMMARY:
Study of BCG Vaccination scars of under five years old children . Estimation of the frequency of children without BCG scar after BCG vaccine . Evaluation of factors which may affect scar formation . Tuberculin skin test response in children without BCG scar . Frequency of vaccine adverse effects as injection-site abscess, lymphadenitis, severe local reaction, and disseminated BCG infection.

DETAILED DESCRIPTION:
Tuberculosis (TB) is an ancient disease, with evidence of skeletal TB found in mummies in both the Old and New World. The causative agent is Mycobacterium tuberculosis, a fastidious, aerobic, acid-fast bacillus Tuberculosis (TB) remains a major global health problem. It ranks as the second leading cause of death from an infectious disease worldwide, after the human immunodeficiency virus (HIV). The latest estimates by the World Health Organization (WHO) reported that there were 9 million new cases in 2011 and 1.4 million TB deaths . Moreover, it is one of the top 10 causes of global mortality and affects low-income countries in particular. About half a million children (0-14 years old) are ill with TB, and 64,000 children died from the disease in 2011 . In Egypt, TB is considered the third most important public health problem after schistosomiasis and hepatitis C .

TB in children is often missed or overlooked due to non-specific symptoms and difficulties in diagnosis. This has made it difficult to assess the actual magnitude of the childhood TB epidemic, which may be higher than currently estimated.

There is an urgent need for public attention, prioritisation, commitment and funding for this disease that today should never take the life of a child.

Bacillus Calmette-Guérin (BCG) vaccine : a live attenuated vaccine that has been in use since 1921, is the most widely used vaccine worldwide . BCG is efficacious against the most severe forms of tuberculosis (TB) such as tuberculosis meningitis (73% protection) and miliary TB (77% protection) in children younger than 5 years .

It is one of the mandatory vaccines recommended by the ministry of health(MOH) of Egypt.

BCG vaccination became compulsory in all governorates of Egypt since 1974 . the recommended schedule of BCG is eight weeks postnatal. The usual response to administer BCG vaccine is the development of erythema or a papule at around 2 weeks, followed by an ulcer and healing with a scar at 6 weeks at the site of the injection.

Although the size of reaction after vaccination is not generally thought to influence the degree of protection offered by BCG, the presence of the BCG scar has been used as a criterion to assess the uptake of vaccination .

However, the sensitivity of BCG scar as an index of vaccination status is still the subject of controversy. Failure to form scar may be related to factors such as lack of maturation of the immune system, faulty technique or unipotent vaccine.

Adverse effects of Bcg vaccine: were classified, according to World Health Organization definitions , as injection-site abscess, lymphadenitis, severe local reaction, and disseminated BCG infection.

Tuberculin skin test response:

The reaction is read by measuring the diameter of induration (palpable raised, hardened area) across the forearm (perpendicular to the long axis) in millimeters. If there is no induration, the result should be recorded as "0 mm". Erythema (redness) should not be measured.

* 5 mm or more is positive in
* An HIV-positive person
* Persons with recent contacts with a TB patient
* Persons with nodular or fibrotic changes on chest X-ray consistent with old healed TB
* Patients with organ transplants, and other immunosuppressed patients
* 10 mm or more is positive in
* Recent arrivals (less than five years) from high-prevalence countries
* Injection drug users
* Residents and employees of high-risk congregate settings (e.g., prisons, nursing homes, hospitals, homeless shelters, etc.)
* Mycobacteriology lab personnel
* Persons with clinical conditions that place them at high risk (e.g., diabetes, prolonged corticosteroid therapy, leukemia, end-stage renal disease, chronic malabsorption syndromes, low body weight, etc.)
* Children less than four years of age, or children and adolescents exposed to adults in high-risk categories
* 15 mm or more is positive in
* Persons with no known risk factors for TB.

the study aims to• Estimate the frequency of children without BCG scar after bcg vaccination.

* Evaluate factors which may affect scar formation.
* Tuberculin skin test response in children without BCG scars if indicated.
* Frequency of vaccine adverse effects

Exclusion criteria:

* Infants with skin lesion on the left forearm.
* Infant treated with steroids or intravenous immune globulins.
* Infants with immunodeficiency.
* Severe sepsis.
* Infants with congenital anomalies.

All cases included in the study will be subjected to

* Full clinical history including: Birth weight, nutritional status, gender, gestational age, weight at time of vaccination, mother awareness.
* Detailed clinical examination: including site of bcg scar.
* Tuberculin test in negative BCG scar children.
* Revaccination of negative BCG scar children.

ELIGIBILITY:
Inclusion Criteria:

- Children between 6 and 60 months of age.

Exclusion Criteria:

* • Infants with skin lesion on the left forearm.

  * Infant treated with steroids or intravenous immune globulins.
  * Infants with immunodeficiency and malnutrition.
  * Severe sepsis.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
number of children without bcg scar after bcg vaccination and factors that may lead to that nummber of children with adverse effects from bcg vaccine using clinical data about children included in the study | one year
  bcg vaccination reaction and adverse effects and factors affecting scar formation

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ghazaly, professor, Principal Investigator — assiut universitypediatric hospital; mustafa embaby, assistprof, Principal Investigator — assiut universitypediatric hospital